CLINICAL TRIAL: NCT06379776
Title: Classification of Thoracic and Lumbar Spinal Fractures. Development of an Interactive 3D Model for Pedagogy.
Brief Title: 3D Model - Classification of Thoracic and Lumbar Spinal Fractures.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Paris-Sud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LabForSIMS-LC1
Record Dates: First submitted 2024-01-16; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Spine Disease
Keywords: simulation; surgery; 3D model
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D model group (Experimental): Residents having access to the 3D model
  Interventions: Other: Education through a 3D model
- Traditional teaching group (Active Comparator): Residents having access to traditional educational support
  Interventions: Other: Education through a traditional pedagogical support

INTERVENTIONS:
Other: Education through a 3D model — Training through a 3D model of the spine fractures
  Arms: 3D model group
Other: Education through a traditional pedagogical support — Training through a traditional pedagogical support
  Arms: Traditional teaching group

SUMMARY:
The goal of this clinical trial is to evaluate and compare the effectiveness of a 3D interactive model versus traditional teaching methods in enhancing the teaching of thoracic and lumbar spine fractures classification (AO Spine) among orthopedic residents.

The main questions this study aims to answer are:

Does the use of a 3D interactive model improve residents' knowledge regarding the AO Spine classification of spine fractures compared to traditional teaching methods? To what extent does the utilization of a 3D interactive model enhance understanding of spinal anatomy, injury mechanisms, pathophysiology, and fracture diagnosis among surgical residents?

Participants will be randomly assigned to either:

Group A: Access to the 3D interactive model depicting thoracic and lumbar spine fractures based on the AO Spine classification. They can explore fractures, access textual information, and anatomical annotations.

Group B: Traditional teaching materials including slides, texts, and diagrams illustrating spine fractures according to the AO Spine classification.

Researchers will compare the post-training knowledge and confidence levels in managing spine fractures between the two groups to assess the efficacy of the 3D model.

Participants will be required to fill out pre- and post-training questionnaires assessing their knowledge, experience with 3D educational tools, confidence levels in managing spine fractures, and satisfaction with the teaching method.

The study aims to ascertain if the use of the 3D model significantly enhances residents' comprehension of spine fractures compared to conventional teaching methods within the orthopedic curriculum.

DETAILED DESCRIPTION:
Detailed Study Protocol

Primary Study - Validation of 3D Interactive Model for Teaching AO Spine Classification for Thoracic and Lumbar Spine Fractures

Introduction:

Thoracic and lumbar spinal fractures are common in orthopedic and trauma surgery. Despite various classifications available, such as the AO Spine classification, understanding these fractures, especially for novice residents, can be challenging. In response, a 3D interactive model has been developed to support the classification teaching. A preliminary validation study with expert surgeons has been conducted.

Objectives:

This study aims to validate the effectiveness of a 3D model in teaching thoracic and lumbar spine fractures compared to traditional teaching methods. The primary objective is to assess whether the use of the 3D model improves residents' knowledge regarding AO Spine classification, anatomy, injury mechanisms, pathophysiology, and diagnosis of spine fractures.

Methods:

This prospective randomized validation study will start in May 2024.

* 3D Model Design and Validation: The pedagogical 3D model was created using Blender® software. Validation, in terms of anatomical realism and adherence to AO Spine classification, was performed through a pilot study involving 24 expert spine surgeons.
* Participant Selection: Sixty orthopedic residents nationwide will be recruited. Sample size determination considered resource availability and study duration.
* Study Protocol: Data collection will involve questionnaires assessing pre-training knowledge, experience with 3D tools, confidence levels in managing spine fractures, and post-training assessments. Residents will be randomized into two groups: 3D model group (Group A) and traditional teaching group (Group B).
* Statistical Analysis: Data analysis will utilize Stata version 16.0. Descriptive statistics and comparative analyses will be employed, considering a significance level of p < 0.05.
* Ethics: Informed consent will be obtained. Data will be anonymized, stored securely. Data handling will comply with privacy regulations. At the end of the study, all interns will access both teaching supports.

Two additional studies will be conducted as follows, with the same protocol :

1. 3D screen-based simulator of a complete Transforaminal Interbody Lumbar Fusion (TLIF) surgical procedure
2. Comparison between Virtual Reality and Screen-based simulators for Transforaminal Interbody Lumbar Fusion (TLIF) surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Residents entering residency in Orthopaedic Surgery for the first study on AO Spine classification of thoracolumbar fractures
* Any resident in Orthopaedic Surgery (from 1st year to 6th year) for the second and third study on TLIF surgical simulation
* Written informed consent

Exclusion Criteria:

* Any prior experience in spine surgery for the 1st year residents for the first study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-25 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Specific Questionnaire | Immediately after the intervention
  The primary outcome measure will be the final score on the post-test questionnaire assessing the student's knowledge. Each of the three studies will have specific questionnaire.

SECONDARY OUTCOMES:
Objective Structured Assessment of Technical Skills (OSATS) | Immediately after the intervention
  Assessment questionnaire of the students technical skills during the validation phase on sawbones. OSATS scale ranges from 7 to 35 points: the higher the score, the better the technical surgical skills.
Subjective questionnaire | Immediately after the intervention
  Final score on a subjective questionnaire evaluating ease of use, immersion and satisfaction with the simulator. Each item ranges from 1 to 10, 10 being the best score (easiest use of the simulator, best immersion, best satisfaction).

IPD SHARING:
Plan to Share IPD: Yes
IPD can be made available on reasonable request
Supporting Information: Study Protocol, SAP